CLINICAL TRIAL: NCT00489788
Title: MRI Assessment of Right and Left Ventricular Strain, Associated Function, Volume and ECG Parameters as Predictors of Optimal Timing for Pulmonary Valve Replacement in Patients Post Repair for Tetralogy of Fallot
Brief Title: Predictors for Pulmonary Valve Replacement - Anatomic and Hemodynamic Using MRI
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, W. James Parks, MD, Principal Investigator, Emory University
Other Study IDs: IRB00000990
Record Dates: First submitted 2007-06-19; First posted 2007-06-21 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Congenital Disorders
Keywords: MRI; Ventricular Strain; Pulmonary Valve Replacement; Post Tetralogy of Fallot
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Magnetic Resonance Imaging (MRI) is a non-invasive test that can look at the heart without using radiation. An MRI will allow the doctors to look at the heart in order to assess how well the ventricle is pumping, the amount of blood that it is pumping in addition to how much it is stretching. An engineer at Georgia Tech has developed a new way of looking at an MRI. It is believed that this new way of looking at an MRI may be better able to tell us when to replace the valve in these children. If this new process works, not only can we apply it now but we will be able to look at previously performed MRIs and gather more information about these children and their heart function in order to help these and other children in the future.

We are planning on enrolling 30 subjects in this study. Some of the subjects will be enrolled and have their MRI strictly for the purpose of this study. Some of the subjects will be already scheduled for a routine MRI of their heart and we will ask them if we can do extra images for the study while they are already here.

DETAILED DESCRIPTION:
Cardiovascular disease remains a leading cause of morbidity and death in the Western World. Assessment of Myocardial function has proven to be a clinically relevant method for monitoring and evaluating outcomes of medical therapy and surgery for structural lesions or acquired disease.

Tetralogy of Fallot (TOF) is the most common form of cyanotic congenital heart disease with a prevalence of 0.26 to 0.8 per 1000 live births The current surgical approach favors primary repair in infancy. This decreases the necessity for palliative procedures and has a low operative mortality. Complete repair often results in pulmonary regurgitation (PR), which is generally well tolerated in infancy. Late complications may include ventricular dilatation, tricuspid regurgitation, diastolic and systolic dysfunction, arrhythmias and sudden cardiac death.

Pulmonary valve replacement (PVR) is required in approximately 20% of patients with repaired TOF and has a 1-4% peri-operative mortality. Thus, early intervention may reduce irreversible right ventricle injury; however no definitive tools are presently available for determining patients at risk.

Myocardial strain analysis has not been critically evaluated to determine its value for predicting RV failure. This study will investigate the practicality and accuracy of a novel mathematical method, developed by the investigators, for analysis of cardiac deformation recovery from dynamic Cardiovascular Magnetic Resonance Imaging (CMRI) sequences. The proposed method requires structural MRI data, offering several important advantages over existing methods. These include reduced requirements in imaging time and analysis effort, and the option to use a large database of prior structural MRI studies of TOF patients in retrospective research.

This three-dimensional method is mathematically based on nearly incompressible tissue deformations. The project proposes validation of technique, comparing its results with current 'gold standard' methods that presently use CMRI myocardial tagging and phase velocity mapping, as a pilot study for clinical validation of strain imaging in TOF patients. The method tracks movement of myocardial tissue throughout the cardiac cycle to compute strain associated with normal and a clinical disease state.

During the study we will customize the method and software for specific use with CMRI and TOF. We will test the method on normal controls and TOF patients pre and post pulmonary valve replacement.

ELIGIBILITY:
Inclusion Criteria:

* Thirty (30) patients diagnosed with Tetralogy of Fallot.
* Ten (10) patients with previously repaired post-PVR.
* Ten (10) normal control subjects.
* Meet the eligibility criteria for MRI.
* Age range: 3-30 years
* Informed consent being obtained from the legal guardians and/or patients.

Exclusion Criteria:

* Outside target age range.
* Contra-indications to MRI such as metallic implants
* Acquired (non-congenital) heart disease

Ages: 3 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pediatrics and young adults aged 3-30 years following surgical repair of Tetralogy of Fallot. Also looking at normal control subjects.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2008-09; Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: W.James Parks, MD, Principal Investigator — Emory University